CLINICAL TRIAL: NCT04146311
Title: Effect of Short-term Motor Training on Accuracy and Precision of Knee Movement in Human With and Without Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Kelun Wang, Associate professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20170080
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Isotonic Saline; Hypertonic Saline; Healthy Eld Human; Knee Pain Chronic
MeSH Terms: interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypertonic saline (Active Comparator): A bolus injection (0.25 ml) of hypertonic saline (5%) is injected into the left infrapatellar fat pad.
  Interventions: Drug: Hypertonic saline; Other: Motor training
- Isotonic saline (Placebo Comparator): A bolus injection (0.25 ml) of isotonic saline (0.9 %) is injected into the left infrapatellar fat pad.
  Interventions: Drug: isotonic saline; Other: Motor training
- Motor training (Experimental): All the subjects recruited need to have a short-term motor task training at home. 30 times a session, totally 2 sessions a day for 6 days
  Interventions: Other: Motor training

INTERVENTIONS:
Drug: Hypertonic saline — A bolus injection (0.25 ml) of hypertonic saline (5%) into the left infrapatellar fat pad.
  Arms: Hypertonic saline
Drug: isotonic saline — A bolus injection (0.25 ml) of isotonic saline (5%) into the left infrapatellar fat pad.
  Arms: Isotonic saline
Other: Motor training — All the subjects recruited need to have a short-term motor task training at home. 30 times a session, totally 2 sessions a day for 6 days

SUMMARY:
The objects of this research are to investigate the ability of the motor learning and test the possible differences between younger and older healthy human, and between non-pain and acute experimental pain and chronic clinical pain conditions.

DETAILED DESCRIPTION:
The project consists of four experimental studies. In the first experiment, younger and older healthy human subjects are involved in a short-term neuromuscular training on the accuracy and precision of knee movement to investigate the possible age effect of the motor learning. The second experiment focuses on the experimental pain on the learning effect of the younger subjects. The third experiment will investigate a group of knee osteoarthritis patients to show the influence of chronic pain on the motor training compared with age-, gender-matched pain free subjects. 3D camera tracking system will be used to record the knee movements at the baseline and after 6-day motor task training. The variability in amplitude of the values of knee movements was transformed to percentage in relation to the target position (accuracy) or to the mean position (precision). The results of the study will contribute to both basic and clinical understanding of the mechanisms related to knee movement control and influences of varies painful conditions.

ELIGIBILITY:
Inclusion Criteria:

* • Aged 18-30 or 50-65 years

  * Free from ongoing or chronic pain
  * Right dominant leg
  * Speak and understand English
  * Aged 50-65 years.
  * Diagnosed with knee OA (according to American College of Rheumatology classification) with pain in left or both knees for more than six months
  * Have ongoing pain rated above 2 on a 0-10 Visual Analogues Scale (VAS) in the previous week.
  * Right dominant leg
  * Speak and understand English
  * Aged 50-65 years
  * Diagnosed with knee OA
  * Have had total knee arthroplasty on left or both knees
  * Right dominant leg
  * Speak and understand English

Exclusion Criteria:

* • Pregnancy or intent to become pregnant, breast feeding

  * Regular use of analgesics, including simple analgesia and NSAIDs
  * Frequent recreational drug or alcohol use
  * History of knee joint pathology or injury
  * Previous neurologic, musculoskeletal or mental illnesses
  * Practicing sport activities on a regular basis
  * Lack of ability to cooperate
  * Regular use of analgesics, including analgesia and NSAIDs for the last 24 hours
  * Frequent recreational drug or alcohol use
  * Previous neurologic, musculoskeletal or mental illnesses
  * Practicing sports activities on a regular basis
  * Lack of ability to cooperate
  * Regular use of analgesics, including analgesia and NSAIDs for the last 24 hours
  * Frequent recreational drug or alcohol use
  * Other disorders or injuries in the knee joints
  * Previous neurologic, musculoskeletal or mental illnesses
  * Practicing sports activities on a regular basis
  * Lack of ability to cooperate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
knee movement assessment | Change from baseline, up to 7 days after the first session
  There are two sessions in total, seperated by a 6 days motor training. Using 3D camera to calculate the accuracy and precision of knee movements at 30, 45, 60 degree respectively both with and without visual feedback (baseline), before and after motor training, also before and after injection.

SECONDARY OUTCOMES:
Assessment of pain | Only on day 7 (second session), up to 24 hours
  Immediately following the injection, participants will be instructed to rate the pain intensity for ten minutes using a digital visual analogue scale (VAS; eVas Software: Aalborg University, Denmark), on a tablet.The scale will be measured from 0 to10, where 0 represents 'no pain' and 10 represents 'worst pain imaginable'.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark

REFERENCES:
- [Derived] Liao S, Arendt-Nielsen L, Wang K, Hirata RP. Effect of Experimental Pain and Visual Feedback on the Accuracy and Precision of Knee Joint Position Sense. Pain Res Manag. 2025 Apr 10;2025:9328803. doi: 10.1155/prm/9328803. eCollection 2025. PMID 40255927